CLINICAL TRIAL: NCT04650672
Title: Daily Testing at Home by NV-AMD Subjects With Notal Home OCT.
Status: Completed | Type: Observational
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2020.004
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Retinal Neovascularization
Keywords: AMD self-scanning Home-OCT
MeSH Terms: conditions — Retinal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the ability of subjects with NV-AMD to perform sequential daily self-imaging of their eyes with the self-operated Notal Home OCT device in their homes for 90 days without on-site supervision. The study will include up to 15 subjects.

DETAILED DESCRIPTION:
Office Visit screening visit:

1. The patient will be informed concerning the study and sign the Informed Consent Form (ICF) prior to conduct of any study procedures
2. The following data will be collected for each study subject:

   a .Subject's DOB (if allowed) or age b. Gender c .Race d. Ethnicity
3. BCVA on both eyes on the day of the visit
4. Both eyes of the subject will be scanned, non-dilated, with either a commercial Zeiss Cirrus or Heidelberg Engineering Spectralis OCT device with one (1) acceptable volume scan of each eye being obtained
5. Both eyes of the subject that meet all screening criteria will be enrolled
6. The following data will be collected for the study eye(s):

   1. Qualifying diagnosis for the study eye from the subject's medical record
   2. From the subject's medical record, the presence of other ophthalmic conditions including but not limited to:

   i. Cataract ii. Glaucoma iii. Dry Eye iv. Other macula findings
7. The subject will receive a general overview of the self-operation of the Notal Home OCT at the investigational clinic facility by trained study personnel. A Notal Home OCT device is then assigned to the subject.
8. The subject will be reminded that the Notal Home OCT will be delivered to their home and instructed to self-image the study eye(s) daily using a Notal Home OCT device at home for 90 days.

Home Set-up with Remote Assistance (Day 0)

Following confirmation of subject eligibility at the Enrollment visit and the subject is enrolled in the study:

1. The subject will be contacted by the NVDC to verify their delivery address.
2. The device will be delivered to the subject's home, with confirmation sent back to the NVDC.
3. Remote support is available by the NVDC via phone during standard business hours of 8am - 6pm EST, if needed.
4. The subject will follow the steps detailed in the Set-up Guide included in the box

In-Home Phase (Day 0 to Day 90) Following set-up of the Notal Home OCT,

1. Day 0: The subject will review the tutorial and will perform one calibration session for each eye.
2. Day 1: The subject will perform the first self-imaging session with the Notal Home OCT on both eyes followed by automated transmission of the scans. This first session will be considered a practice session.
3. Days 2-90: The patient will perform one self-imaging session followed by automated transmission on both eyes at home with the Notal Home OCT each day.

If an eye cannot calibrate during 5 separate attempts or fails to test 5 consecutive times, the subject will be notified by the NVDC to discontinue self-imaging this eye. If there is a fellow eye also enrolled in the study, the fellow eye will continue

Weekly Review of Notal Home OCT Images by the PI:

The physician will review patient images on a weekly basis to perform an assessment of daily fluid status and document their observations in the CRF.

Routine Care Visits:

Routine care visits may be conducted at the investigator's discretion. The following procedures will be performed at the routine care visits: BCVA, Spectralis or Cirrus OCT, 3. Initiate treatment, if necessary, and document which anti-VEGF drug is used.

At Office Exit Visit (approximately 90 days after Day 0)

Subjects will return to the clinic for an office visit approximately ninety (90) days after the Day 0 (Home Set-up) Visit. At this visit, the exams will be conducted in the following order:

1. BCVA will be performed on both eyes.
2. Both eyes of the subject will be imaged, using a Cirrus or Spectralis OCT, and reviewed by the PI to determine fluid status.
3. Initiate standard of care and treatment, if necessary.
4. Collect AEs, if applicable.
5. Subject completes the Notal Home OCT Subject User Questionnaire.
6. Exit subject from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to speak and understand English with fluency.
2. Ability to understand and agree to contents of informed consent either in writing or verbally.
3. At least 55 years of age on date of Screening Visit.
4. Diagnosed with NV-AMD in at least one eye and initiation of anti-VEGF treatment in that eye.
5. At least one enrolled eye per subject had retinal fluid treated with anti-VEGF in the prior 6 months, with a treatment interval of 8 weeks or less.
6. Visual Acuity of 20/320 or better.
7. Available and willing to conduct daily self-imaging at home for the duration of the trial.

Exclusion Criteria:

1. Any other retinal disease in the study eye requiring steroidal or anti-VEGF injections (anti-VEGF injections during the study period must be for NV-AMD).
2. Subject's schedule not conducive to completing daily tests at home with the Notal Home OCT device for the duration of the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include approximately fifteen (15) subjects diagnosed with NV-AMD in at least one eye with initiation of anti-VEGF treatment within the past 6 months, at treatment intervals 8 weeks or less, in the NV-AMD eye. At least 50% of the subjects in each of the two study sites with active NV-AMD at time of enrollment in at least one eye, defined as presence of intra- and/or subretinal fluid as seen on the office OCT. Approximately 50% of the eyes with fluid will have intra retinal fluid and at approximately 50% will have sub retinal fluid. Eyes may have both types of fluid.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of successful imaging attempts during daily testing. | 90 days

SECONDARY OUTCOMES:
Percentage of eyes successfully completed the set up and calibration | 10-15 minutes
Percentage of volume scans with Manufacturer Image quality Index (MSI) >=2 (in a scale of 0-7, where 2 is a pre-defined acceptable-MSI cutoff) | 90 days
Percentage of eligible B-scans out of the maximum 88 in each volume scan during daily testing | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston, Boston, MA.; Nancy Holekamp, MD, Principal Investigator — Pepose Vision Institute, Chesterfield, MO.
Locations (2):
- United States (2):
  - Ophthalmic Cons. of Boston, Boston, Massachusetts
  - Pepose Vision Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided